CLINICAL TRIAL: NCT00211237
Title: A Multicenter, Prospective, Randomized, Controlled Study to Compare Balloon Kyphoplasty to Non-surgical Fracture Management in the Treatment of Painful, Acute Vertebral Body Compression Fractures in Cancer Patients
Brief Title: CAFE Study - Cancer Patient Fracture Evaluation
Acronym: CAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Organization: Medtronic Spinal and Biologics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP0401 - CAFE Study
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2017-06

CONDITIONS: Cancer; Spinal Fractures
Keywords: Balloon Kyphoplasty; Cancer; Vertebral Compression Fracture; Back Pain; Spine
MeSH Terms: conditions — Neoplasms; Spinal Fractures; Back Pain | interventions — Kyphoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balloon Kyphoplasty (BKP) (Experimental): The subjects assigned to this group will undergo the treatment with Balloon kyphoplasty for their painful VCFs.
  Interventions: Device: Balloon Kyphoplasty
- Non Surgical Management (Active Comparator): The subjects in this group will undergo the non-operative treatments aimed at alleviation of back pain and restoration of decreased function associated with VCFs.
  Interventions: Other: Non Surgical Management

INTERVENTIONS:
Device: Balloon Kyphoplasty — Ballon Kyphoplasty is a minimally invasive technique aimed at reduction of VCFs using KyphX® Inflatable Bone Tamps followed by fracture fixation with KyphX® HV-R™ Bone Cement.
  Other Names: KyphX Inflatable Bone Tamps
  Arms: Balloon Kyphoplasty (BKP)
Other: Non Surgical Management — Non-surgical treatment includes, but is not limited to, the following: back brace, pain medication, physical therapy, walking aids, bed rest, and radiation treatment.
  Arms: Non Surgical Management

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of balloon kyphoplasty treatment for painful, acute, vertebral compression fractures (VCFs) as compared to standard non-surgical therapy in patients with cancer.

DETAILED DESCRIPTION:
1. STUDY OBJECTIVES AND ENDPOINTS

1.1. Objectives

The primary objective of this study is to evaluate the safety and effectiveness of balloon kyphoplasty treatment for painful, acute, VCFs as compared to standard non-surgical therapy in patients with cancer.

1.2. Primary Endpoint

The primary endpoint of the study is the improvement in functional status, as measured by the Roland-Morris Disability Questionnaire (RDQ) at 1 month. The primary hypothesis of the study is that the mean improvement will be larger in subjects initially assigned to management with balloon kyphoplasty. Note that all subjects will undergo 12 months of follow-up after initial treatment assignment.

1.3. Secondary Endpoints

The following secondary endpoints will also be examined. Comparisons will be made at each follow-up visit.

Safety:

* Rate of study treatment-related adverse events
* Change in neurological status

Clinical:

* Change in functional status as assessed with Karnofsky Performance Scale
* Change in quality of life as assessed by the SF-36v2™ Health Survey
* Change in back pain, as measured by a 10-point Numerical Rating Scale (NRS)
* Change in back-pain analgesics used
* Change in ambulation status
* Changes in activities of daily living
* Time to treatment failure

Radiographic:

* Change in spinal deformity, defined as the degree of spine angulation as assessed by an independent radiologist at the core laboratory
* Rate of subsequent vertebral body fractures, as assessed by independent radiologists at the core lab

In each case, the study hypothesis is that treatment with balloon kyphoplasty will result in an improvement in clinical or radiographic outcomes compared to baseline and compared to non-surgical treatment, with a preservation of outcomes in long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. One to 3 painful (pain on palpation/percussion over fractured vertebral body) VCF(s), T5-L5, with either bone marrow edema imaged by magnetic resonance imaging (MRI) or a fracture imaged by plain radiographs using the method of Genant
2. Pain NRS score ≥4 on a scale of 0 to 10

   * When the patient is newly diagnosed with multiple myeloma, the pain assessment must not be done until after completion of at least one pulse of steroid therapy or one week after the initiation of active multiple myeloma therapy.
3. Roland Morris Disability Questionnaire score ≥ 10 on a scale of 0 to 24
4. Patients must be at least 21 years old.
5. No change in chemotherapy regimen (change in dose(s) permitted) for 1 month prior to enrollment
6. No change in chemotherapy regimen (change in dose(s) permitted) planned for at least 1 month following enrollment
7. No major surgery to the spine planned for at least 1 month following enrollment
8. Life expectancy of ≥ 3 months
9. Patient has sufficient mental capacity to comply with the protocol requirements
10. Patient has stated availability for all study visits
11. Patient is able to understand the risks and benefits of participating in the study and is willing to provide written informed consent.

Exclusion Criteria:

1. Patients with primary tumors of the bone (e.g., osteosarcoma) or solitary plasmacytoma at site of the index VCF. Patients with these tumors in anatomic sites other than the index VCF are eligible.
2. Concurrent Phase I investigational anti-cancer treatment
3. Significant clinical morbidities (aside from the index fracture(s) and cancer) that may potentially interfere with the collection of data concerning pain and function
4. VCF morphology deemed unsuitable for balloon kyphoplasty
5. Additional non-kyphoplasty surgical treatment is required for the index fracture
6. Patients requiring the use of high-dose steroid (≥ 100 mg prednisone or 20 mg dexamethasone per day), intravenous (IV) pain medication, or nerve block to control chronic back pain unrelated to index VCF(s). Patients who receive high-dose steroids for treatment of their cancer (for at least 30 days) are eligible.
7. Patients with a platelet count of < 20,000 measured at the time of hospital admission for the procedure
8. Spinal cord compression or canal compromise requiring decompression
9. Patients with osteoblastic tumors at the site of index VCF. Patients with osteoblastic tumors outside of vertebral levels intended for kyphoplasty may be enrolled.
10. Medical/surgical conditions contrary to the balloon kyphoplasty procedure (e.g., in the presence of active or incompletely treated local infection)
11. Known allergy to bone cement or contrast medium used in the treatment of study subjects
12. MRI contraindication (e.g., cerebral aneurysm clips, pacemaker, implanted biostimulators, cochlear implants, penile prosthesis)
13. Positive baseline pregnancy test (for women of child-bearing potential)
14. Patients who may require allogeneic bone marrow transplantation during the course of the study.

Other Reasons for Lack of Enrollment:

A. Patient is afraid to have surgery

B. Patient is afraid to have anesthesia

C. Patient/family is not willing to participate in research

D. Patient is not willing to be randomized

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2005-05; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Berenson, M.D., Principal Investigator — Institute for Myeloma & Bone Cancer Research; Frank Vrionis, M.D., Principal Investigator — H. Lee Moffitt Cancer Center
Locations (20):
- United States (9):
  - Valley Radiology Inc., UCSD, Escondido, California
  - Boulder Neurosurgical Associates, Boulder, Colorado
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Sibley Memorial Hospital, Chevy Chase, Maryland
  - Greater Oncology Associates, Silver Spring, Maryland
  - Karmanos Cancer Center, Detroit, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (2):
  - St. Vincent's Hospital, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Institut Jules Bordet, Brussels, Belgium
- Canada (3):
  - Foothills Hospital, Calgary, Alberta
  - Toronto Western Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
- Germany (2):
  - Charité Virchow-Klinikum, Berlin
  - Medizinische Hochschule, Hanover
- National Center for Spinal Disorders, Budapest, Hungary
- Akademiska Sjukhuset, Uppsala, Sweden
- Royal London, London, United Kingdom

REFERENCES:
- [Derived] Berenson J, Pflugmacher R, Jarzem P, Zonder J, Schechtman K, Tillman JB, Bastian L, Ashraf T, Vrionis F; Cancer Patient Fracture Evaluation (CAFE) Investigators. Balloon kyphoplasty versus non-surgical fracture management for treatment of painful vertebral body compression fractures in patients with cancer: a multicentre, randomised controlled trial. Lancet Oncol. 2011 Mar;12(3):225-35. doi: 10.1016/S1470-2045(11)70008-0. Epub 2011 Feb 16. PMID 21333599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 134 enrolled subjects, 70 were randomized to Balloon Kyphoplasty and 64 to non-surgical management (NSM). Two of the subjects who were randomized to Balloon Kyphoplasty and 3 of the subjects who were randomized to NSM were excluded from the mITT and PP Populations, because they terminated in a few days of enrolment and had no treatment.
Pre-assignment Details: Crossover from the NSM group to Balloon Kyphoplasty group was permitted after completion of the 1-month evaluation.
Groups:
- Balloon Kyphoplasty: The subjects assigned to this group have undergone the treatment with Balloon Kyphoplasty for their painful VCFs.
- Non-surgical Management: The subjects in this group have undergone the non-operative treatments aimed at alleviation of back pain and restoration of decreased function associated with VCFs.
- Crossover: Subjects in this group were randomized to NSM, then, crossed over to Balloon Kyphoplasty after completion of the 1-month evaluation in NSM group.
Period: Baseline
Arm/Group | Balloon Kyphoplasty | Non-surgical Management | Crossover
Started | 70 | 64 | 0
Completed | 68 | 61 | 0
Not Completed | 2 | 3 | 0
Not completed — Withdrew | 1 | 3 | 0
Not completed — Refused random assignment | 1 | 0 | 0
Period: 1 Month
Arm/Group | Balloon Kyphoplasty | Non-surgical Management | Crossover
Started | 68 | 61 | 0
Completed | 65 | 52 | 0
Not Completed | 3 | 9 | 0
Not completed — Death | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrew | 0 | 4 | 0
Not completed — Additional surgery needed | 1 | 0 | 0
Not completed — Non-medical problem | 0 | 2 | 0
Period: 3 Months
Arm/Group | Balloon Kyphoplasty | Non-surgical Management | Crossover
Started | 65 | 18 (34 patients crossed over to Balloon Kyphoplasty.) | 34
Completed | 57 | 14 | 33
Not Completed | 8 | 4 | 1
Not completed — Death | 7 | 3 | 0
Not completed — Could not comply with protocol | 1 | 0 | 0
Not completed — Withdrew | 0 | 1 | 0
Not completed — Non-medical problem | 0 | 0 | 1
Period: 6 Months
Arm/Group | Balloon Kyphoplasty | Non-surgical Management | Crossover
Started | 57 | 11 (3 patients crossed over Balloon Kyphoplasty) | 36
Completed | 49 | 9 | 33
Not Completed | 8 | 2 | 3
Not completed — Death | 6 | 0 | 3
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Could not comply with protocol | 0 | 2 | 0
Period: 12 Months
Arm/Group | Balloon Kyphoplasty | Non-surgical Management | Crossover
Started | 49 | 8 (1 patient crossed over Balloon Kyphoplasty) | 34
Completed | 40 | 6 | 28
Not Completed | 9 | 2 | 6
Not completed — Death | 8 | 2 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrew | 0 | 0 | 1
Not completed — unrelated medical problem | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Non Surgical Management: The subjects in this group have undergone the non-operative treatments aimed at alleviation of back pain and restoration of decreased function associated with VCFs.
- Total: Total of all reporting groups
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Total
Number analyzed (Participants) | 70 | 64 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.8) | 63.0 (11.4) | 63.9 (11.0)
Sex/Gender, Customized [Number; unit: participants]
  Male | 28 | 26 | 54
  Female | 40 | 35 | 75
  Missing | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Functional Status, as Measured by the Roland-Morris Disability Questionnaire (RDQ) at 1 Month
Description: The full scale name is the Roland-Morris Disability Questionnaire; it is a validated measure of physical disability due to back pain.
  The best score is 0 (no disability) and worst is 24 (maximum disability)
Time Frame: Baseline and 1 Month
Population: The analyses of change from Baseline included only patients in the modified Intent-to-Treat (mITT) population who provided evaluable data at both Baseline and at 1 month after receipt of the initially assigned study treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Balloon Kyphoplasty: The subjects assigned to this group received the treatment with Balloon Kyphoplasty for their painful VCFs.
- Non Surgical Management: The subjects in this group received the non-operative treatments that aimed at alleviation of back pain and restoration of decreased function associated with VCFs.
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 63 | 50
score on a scale
  Baseline | 17.6 [16.6 to 18.5] | 18.2 [17.4 to 19.0]
  One month | 9.1 [7.4 to 10.9] | 18.0 [16.9 to 19.0]
  Change from baseline to one month | -8.3 [-10.2 to -6.4] | 0.1 [-0.8 to 1.0]

2. Secondary Outcome: Change in Roland-Morris Disability Questionnaire Score
Description: Roland-Morris Disability Questionnaire (RMDQ) was used to assess the physical disability due to back pain. The best score is 0 (no disability) and worst is 24 (maximum disability).
Time Frame: Baseline, 1 month, 3 months, 6 months, and 12 months
Population: The analysis population was per-protocol analysis, which was based on the treatment that subjects received. Of 61 subjects randomized into NSM group, 38 subjects crossed over from NSM to Kyphoplasty after the 1-month visit, and 23 subjects remained in NSM group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty | Non-Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
units on a scale
  RMDQ score at baseline | 17.6 (3.9) | 17.9 (4.2) | 18.3 (2.6)
  Change from baseline to 1 months: number analyzed (Participants) | 63 | 12 | 38
  Change from baseline to 1 months | -8.3 (7.6) | 0.3 (3.1) | -7.3 (6.8)
  Change from baseline to 3 months: number analyzed (Participants) | 55 | 10 | 36
  Change from baseline to 3 months | -8.9 (7.0) | -2.7 (6.1) | -10.2 (6.1)
  Change from baseline to 6 months: number analyzed (Participants) | 49 | 8 | 33
  Change from baseline to 6 months | -8.2 (6.0) | -3.6 (9.4) | -10.8 (6.1)
  Change from baseline to 12 months: number analyzed (Participants) | 40 | 6 | 27
  Change from baseline to 12 months | -9.7 (6.4) | -4.5 (11.4) | -10.4 (6.0)

3. Secondary Outcome: Change in Functional Status Assessed With the Karnofsky Performance Scale
Description: The Karnofsky Performance Scale rates a patient on an 11-step scale from 0 (dead) to 100 (normal, no complaints, no evidence of disease).
Time Frame: Baseline and 1 month
Population: Subjects were analyzed in modified Intent-to-Treat (mITT) population, based on their randomized treatment group (regardless of crossover). This analysis included all subjects in the mITT population who provided evaluable data at both baseline and 1 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
units on a scale
  Baseline score: number analyzed (Participants) | 68 | 59
  Baseline score | 57.1 (18.0) | 57.3 (15.8)
  Score at 1 month: number analyzed (Participants) | 63 | 49
  Score at 1 month | 73.2 (15.5) | 58.6 (16.2)
  Change from baseline to one month: number analyzed (Participants) | 63 | 49
  Change from baseline to one month | 15.9 (21.2) | 0.6 (11.6)

4. Secondary Outcome: Change in Functional Status Assessed With the Karnofsky Performance Scale
Description: as for outcome 3
Time Frame: Baseline, 1 month, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
units on a scale
  Baseline score: number analyzed (Participants) | 68 | 22 | 38
  Baseline score | 57.1 (18.0) | 55.0 (17.7) | 58.7 (14.6)
  Change from baseline to 1 month: number analyzed (Participants) | 63 | 12 | 37
  Change from baseline to 1 month | 15.9 (21.2) | 0.0 (14.1) | 19.2 (20.6)
  Change from baseline to 3 months: number analyzed (Participants) | 54 | 10 | 36
  Change from baseline to 3 months | 18.0 (23.8) | 10.0 (16.3) | 21.1 (19.1)
  Change from baseline to 6 months: number analyzed (Participants) | 49 | 8 | 33
  Change from baseline to 6 months | 18.0 (23.1) | 12.5 (21.2) | 23.3 (19.8)
  Change from baseline to 12 months: number analyzed (Participants) | 40 | 6 | 27
  Change from baseline to 12 months | 23.0 (25.2) | 21.7 (23.2) | 22.2 (18.0)

5. Secondary Outcome: Change in Back Pain
Description: Back pain was assessed on a 10-point Numerical Rating Scale (NRS) from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline and 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
units on a scale
  Baseline: number analyzed (Participants) | 68 | 60
  Baseline | 7.3 (1.6) | 7.3 (1.4)
  1 month: number analyzed (Participants) | 64 | 50
  1 month | 3.3 (2.8) | 6.9 (1.5)
  Change from baseline to 1 month: number analyzed (Participants) | 64 | 50
  Change from baseline to 1 month | -3.9 (3.2) | -0.6 (1.8)

6. Secondary Outcome: Change in Back Pain
Description: Back pain was assessed on a NRS from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, 1 month, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
units on a scale
  Back pain at baseline | 7.3 (1.6) | 6.8 (1.5) | 7.6 (1.4)
  Change from baseline to 7 days: number analyzed (Participants) | 63 | 16 | 38
  Change from baseline to 7 days | -3.8 (3.0) | -0.7 (1.8) | -4.0 (3.1)
  Change from baseline to 1 month: number analyzed (Participants) | 64 | 12 | 38
  Change from baseline to 1 month | -3.9 (3.2) | -0.9 (2.0) | -4.1 (2.9)
  Change from baseline to 3 months: number analyzed (Participants) | 53 | 10 | 36
  Change from baseline to 3 months | -3.6 (3.3) | -2.1 (2.1) | -4.3 (2.8)
  Change from baseline to 6 months: number analyzed (Participants) | 49 | 8 | 33
  Change from baseline to 6 months | -3.7 (3.2) | -2.4 (3.9) | -4.8 (2.9)
  Change from baseline to 12 months: number analyzed (Participants) | 40 | 6 | 27
  Change from baseline to 12 months | -3.9 (3.2) | -3.0 (3.2) | -4.9 (3.0)

7. Secondary Outcome: Change in Quality of Life.
Description: The SF-36 was used to assess quality of life. The SF-36 results were summarized into two components, a physical component summary score (PCS) (0-100) and a mental component summary score (MCS) (0-100). The higher the score, the better the quality of life.
Time Frame: Baseline and 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
units on a scale
  SF-36 PCS at baseline: number analyzed (Participants) | 68 | 59
  SF-36 PCS at baseline | 25.4 (6.0) | 24.8 (6.4)
  SF-36 PCS at 1 month: number analyzed (Participants) | 58 | 47
  SF-36 PCS at 1 month | 35.2 (10.1) | 26.0 (6.3)
  PCS change from baseline to 1 month: number analyzed (Participants) | 58 | 47
  PCS change from baseline to 1 month | 9.4 (9.4) | 1.0 (6.0)
  SF-36 MCS at baseline: number analyzed (Participants) | 68 | 59
  SF-36 MCS at baseline | 38.2 (13.3) | 37.3 (13.4)
  SF-36 MCS at 1 month: number analyzed (Participants) | 58 | 47
  SF-36 MCS at 1 month | 46.4 (13.0) | 36.1 (13.6)
  MCS change from baseline to 1 month: number analyzed (Participants) | 58 | 47
  MCS change from baseline to 1 month | 9.2 (14.6) | -1.9 (12.7)

8. Secondary Outcome: Change in Quality of Life
Description: The SF-36 were used to assess quality of life. The SF-36 results were summarized into two components, a physical component summary score (PCS) (0-100) and a mental component summary score (MCS) (0-100). The higher the score, the better the quality of life.
Time Frame: Baseline, 1 month, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
units on a scale
  SF-36 PCS at baseline: number analyzed (Participants) | 68 | 22 | 37
  SF-36 PCS at baseline | 25.4 (6.0) | 25.3 (4.8) | 24.5 (7.2)
  PCS change from baseline to 1 months: number analyzed (Participants) | 58 | 11 | 37
  PCS change from baseline to 1 months | 9.4 (9.4) | -0.2 (4.2) | 9.1 (9.5)
  PCS change from baseline to 3 months: number analyzed (Participants) | 52 | 9 | 35
  PCS change from baseline to 3 months | 10.0 (11.1) | 1.1 (6.4) | 11.1 (9.3)
  PCS change from baseline to 6 months: number analyzed (Participants) | 48 | 7 | 32
  PCS change from baseline to 6 months | 9.1 (9.1) | -0.8 (6.2) | 10.8 (9.2)
  PCS change from baseline to 12 months: number analyzed (Participants) | 39 | 5 | 25
  PCS change from baseline to 12 months | 11.7 (10.3) | 1.3 (9.1) | 11.9 (7.9)
  SF-36 MCS at baseline: number analyzed (Participants) | 68 | 22 | 37
  SF-36 MCS at baseline | 38.2 (13.3) | 36.0 (14.7) | 38.1 (12.7)
  MCS change from baseline to 1 month: number analyzed (Participants) | 58 | 11 | 37
  MCS change from baseline to 1 month | 9.2 (14.6) | -1.1 (12.4) | 6.8 (15.9)
  MCS change from baseline to 3 months: number analyzed (Participants) | 52 | 9 | 35
  MCS change from baseline to 3 months | 7.6 (15.0) | 7.3 (13.4) | 9.2 (17.0)
  MCS change from baseline to 6 months: number analyzed (Participants) | 48 | 7 | 32
  MCS change from baseline to 6 months | 8.5 (15.2) | 4.3 (12.1) | 13.1 (15.5)
  MCS change from baseline to 12 months: number analyzed (Participants) | 39 | 5 | 25
  MCS change from baseline to 12 months | 7.8 (15.5) | 5.6 (12.5) | 9.2 (17.1)

9. Secondary Outcome: Change in Activities of Daily Living - Activities Reduced Due to Back Pain in Previous 2 Weeks
Description: The Activities of Daily Living assessment comprised three questions about the effects of back pain or back problems over the previous 2-week period. The patient was asked if they had cut down on usual activities, the number of days in which the patient had cut down on usual activities and the number of days that the patient had spent at least half a day in bed because of back pain or back problems.
Time Frame: Baseline and 1 month
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
percentage of participants
  Activities reduced at baseline | 90 | 97
  No activities reduced at baseline | 8.8 | 1.6
  Don't known at baseline | 1.5 | 0
  Activities reduced at 1 month | 56 | 75
  No activities reduced at 1 month | 38 | 6.6
  Don't know at 1 month | 0 | 0

10. Secondary Outcome: Change in Activities of Daily Living - Activities Reduced Due to Back Pain in Previous 2 Weeks
Description: as for outcome 9
Time Frame: Baseline, 1 month, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
percentage of participants
  Activities reduced at baseline | 90 | 96 | 97
  No activities reduced at baseline | 8.8 | 4.3 | 2.6
  Don't known at baseline | 1.5 | 0 | 0.0
  Activities reduced at 1 month | 56 | 48 | 53
  No activities reduced at 1 month | 38 | 4.3 | 47
  Don't know at 1 month | 0 | 0 | 0
  Activities reduced at 3 months | 37 | 39 | 34
  No activities reduced at 3 months | 43 | 4.3 | 58
  Don't know at 3 months | 0 | 0.0 | 2.6
  Activities reduced at 6 months | 34 | 26 | 32
  No activities reduced at 6 months | 38 | 8.7 | 55
  Don't know at 6 months | 0 | 0 | 0
  Activities reduced at 12 months | 19 | 17 | 39
  No activities reduced at 12 months | 40 | 8.7 | 32
  Don't know at 12 months | 0 | 0 | 0

11. Secondary Outcome: Change in Activities of Daily Living - Number of Days With Reduced Activities Due to Back Pain in Previous 2 Weeks
Description: as for outcome 9
Time Frame: Baseline and 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
days
  Baseline: number analyzed (Participants) | 68 | 60
  Baseline | 10.8 (4.9) | 11.5 (4.3)
  Change from baseline to one month: number analyzed (Participants) | 64 | 50
  Change from baseline to one month | -5.2 (7.1) | 1.1 (4.5)

12. Secondary Outcome: Change in Activities of Daily Living - Number of Days With Reduced Activities Due to Back Pain in Previous 2 Weeks
Description: as for outcome 9
Time Frame: Baseline, 1 month, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
days
  Baseline | 10.8 (4.9) | 12.0 (3.6) | 11.0 (4.8)
  Change from baseline to 1 months: number analyzed (Participants) | 64 | 12 | 38
  Change from baseline to 1 months | -5.2 (7.1) | -0.4 (3.3) | -5.6 (7.2)
  Change from baseline to 3 months: number analyzed (Participants) | 54 | 10 | 36
  Change from baseline to 3 months | -5.5 (7.0) | -1.8 (6.3) | -7.4 (7.1)
  Change from baseline to 6 months: number analyzed (Participants) | 49 | 8 | 33
  Change from baseline to 6 months | -5.0 (7.9) | -2.9 (7.9) | -8.5 (5.2)
  Change from baseline to 12 months: number analyzed (Participants) | 40 | 6 | 27
  Change from baseline to 12 months | -7.8 (6.4) | -5.2 (5.2) | -7.4 (7.3)

13. Secondary Outcome: Change in Activities of Daily Living - Number of Days in Bed Due to Back Pain in Previous 2 Weeks
Description: as for outcome 9
Time Frame: Baseline and 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
days
  Baseline: number analyzed (Participants) | 68 | 60
  Baseline | 6.3 (6.3) | 6.8 (6.0)
  Change from baseline to 1 month: number analyzed (Participants) | 64 | 50
  Change from baseline to 1 month | -4.0 (7.7) | 0.2 (4.7)

14. Secondary Outcome: Change in Activities of Daily Living - Number of Days in Bed Due to Back Pain in Previous 2 Weeks
Description: as for outcome 9
Time Frame: Baseline, 1 month, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
days
  Baseline | 6.3 (6.3) | 8.1 (5.9) | 5.8 (6.0)
  Change from baseline to 1 month: number analyzed (Participants) | 64 | 12 | 38
  Change from baseline to 1 month | -4.0 (7.7) | -0.2 (5.9) | -4.5 (6.0)
  Change from baseline to 3 months: number analyzed (Participants) | 54 | 10 | 36
  Change from baseline to 3 months | -3.4 (7.7) | -4.8 (6.0) | -5.0 (6.1)
  Change from baseline to 6 months: number analyzed (Participants) | 49 | 8 | 33
  Change from baseline to 6 months | -3.8 (7.6) | -4.1 (7.8) | -5.7 (5.9)
  Change from baseline to 12 months: number analyzed (Participants) | 40 | 6 | 27
  Change from baseline to 12 months | -5.8 (6.3) | -4.3 (6.2) | -4.7 (6.8)

15. Secondary Outcome: Ambulatory Status Change From Baseline to One Month
Description: Ambulatory status was assessed using a three-category system, fully ambulatory, ambulatory with assistance, or not ambulatory.
Time Frame: 1 month
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Non Surgical Management: The subjects in this group undergone the non-operative treatments aimed at alleviation of back pain and restoration of decreased function associated with VCFs.
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
percentage of participants
  Fully ambulatory at baseline | 56 | 56
  Assisted ambulatory | 32 | 34
  Not ambulatory | 10 | 8.2
  Ambulatory status improved at 1 month | 16 | 6.6
  No change in ambulatory status at 1 month | 74 | 66
  Ambulatory status worsened at 1 month | 2.9 | 9.8

16. Secondary Outcome: Ambulatory Status Change
Description: as for outcome 15
Time Frame: Baseline, 7 days, 1 month, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
percentage of participants
  Full ambulatory at baseline | 56 | 57 | 55
  Assisted ambulatory at baseline | 32 | 30 | 39
  Not ambulatory at baseline | 10 | 13 | 5.3
  Ambulatory status improved at 7 days | 10 | 0 | 7.9
  Ambulatory status no change at 7 days | 79 | 70 | 87
  Ambulatory status worsened at 7 days | 2.9 | 0 | 5.3
  Ambulatory status improved at 1 month | 16 | 0 | 11
  Ambulatory status no change at 1 month | 74 | 39 | 87
  Ambulatory status worsened at 1 month | 2.9 | 13 | 2.6
  Ambulatory status improved at 3 months | 18 | 4.3 | 16
  Ambulatory status no change at 3 months | 53 | 35 | 76
  Ambulatory status worsened at 3 months | 8.8 | 4.3 | 2.6
  Ambulatory status improved at 6 months | 10 | 4.3 | 16
  Ambulatory status no change at 6 months | 54 | 26 | 63
  Ambulatory status worsened at 6 months | 5.9 | 4.3 | 7.9
  Ambulatory status improved at 12 months | 12 | 4.3 | 16
  Ambulatory status no change at 12 months | 41 | 17 | 53
  Ambulatory status worsened at 12 months | 4.4 | 4.3 | 2.6

17. Secondary Outcome: Index Spinal Deformity Change Measured by Index Vertebral Body Angles From Baseline to 1 Month
Description: Index spinal deformity was measured by Kyphotic angle, local Cobb angle, thoracic and lumbar Cobb angle, and anterior, middle and posterior vertebral body heights for each index VCF.
Time Frame: Baseline and 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
degrees
  Kyphotic angle at baseline: number analyzed (Participants) | 65 | 47
  Kyphotic angle at baseline | 9.523 (8.751) | 10.501 (8.833)
  Kyphotic angle change at 1 month: number analyzed (Participants) | 63 | 47
  Kyphotic angle change at 1 month | 0.135 (5.088) | -0.598 (3.442)
  Thoracic cobb angle at baseline: number analyzed (Participants) | 63 | 46
  Thoracic cobb angle at baseline | 50.976 (17.316) | 51.390 (19.621)
  Thoracic cobb angle change to one month: number analyzed (Participants) | 62 | 46
  Thoracic cobb angle change to one month | 0.666 (9.253) | -0.012 (8.150)
  Lumbar cobb angle at baseline: number analyzed (Participants) | 63 | 46
  Lumbar cobb angle at baseline | -32.335 (16.410) | -33.101 (15.179)
  Lumbar cobb angle change at 1 month: number analyzed (Participants) | 63 | 46
  Lumbar cobb angle change at 1 month | 0.626 (7.075) | 2.883 (7.634)
  Local Cobb angel of T5-L1 at baseline: number analyzed (Participants) | 49 | 40
  Local Cobb angel of T5-L1 at baseline | 22.914 (12.720) | 22.792 (15.191)
  Local cobb angle of T5-L1 change at 1 month: number analyzed (Participants) | 45 | 40
  Local cobb angle of T5-L1 change at 1 month | 1.126 (5.639) | 1.608 (5.631)
  Local cobb angle of L2-L4 at baseline: number analyzed (Participants) | 24 | 22
  Local cobb angle of L2-L4 at baseline | -7.715 (15.470) | -8.291 (14.662)
  Local cobb angle of L2-L4 change at 1 month: number analyzed (Participants) | 23 | 22
  Local cobb angle of L2-L4 change at 1 month | 0.117 (5.694) | -1.149 (5.576)

18. Secondary Outcome: Index Spinal Deformity Change Measured by Index Vertebral Body Angles
Description: as for outcome 17
Time Frame: Baseline, post-operation, 1 month, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
degrees
  Kyphotic angle at baseline: number analyzed (Participants) | 65 | 13 | 36
  Kyphotic angle at baseline | 9.523 (8.751) | 10.806 (8.962) | 11.005 (8.798)
  Kyphotic angle change at post-operation: number analyzed (Participants) | 63 | 23 | 35
  Kyphotic angle change at post-operation | 1.312 (4.909) | NA (NA) — Subjects did not have surgery. | 1.438 (4.191)
  Kyphotic angle change at 1 month: number analyzed (Participants) | 63 | 13 | 35
  Kyphotic angle change at 1 month | 0.135 (5.088) | -0.130 (4.203) | 0.637 (4.545)
  Kyphotic angle change at 12 month: number analyzed (Participants) | 39 | 6 | 28
  Kyphotic angle change at 12 month | 0.954 (5.626) | -1.246 (3.404) | 0.824 (4.425)
  Thoracic cobb angle at baseline: number analyzed (Participants) | 63 | 13 | 35
  Thoracic cobb angle at baseline | 50.976 (17.316) | 53.148 (15.837) | 52.812 (19.671)
  Thoracic cobb angle change at post-op: number analyzed (Participants) | 61 | 23 | 33
  Thoracic cobb angle change at post-op | -1.804 (9.701) | NA (NA) — Subjects did not have surgery. | -2.489 (4.823)
  Thoracic cobb angle change at 1 month: number analyzed (Participants) | 62 | 13 | 36
  Thoracic cobb angle change at 1 month | 0.666 (9.253) | -1.633 (8.212) | -0.457 (5.682)
  Thoracic cobb angle change at 12 months: number analyzed (Participants) | 39 | 6 | 27
  Thoracic cobb angle change at 12 months | 0.988 (8.947) | 0.062 (7.332) | -1.372 (6.187)
  Lumbar cobb angle at baseline: number analyzed (Participants) | 63 | 13 | 34
  Lumbar cobb angle at baseline | -32.335 (16.410) | -31.218 (12.656) | -32.906 (15.718)
  Lumbar cobb angle change at post-op: number analyzed (Participants) | 60 | 23 | 33
  Lumbar cobb angle change at post-op | -0.472 (5.617) | NA (NA) — Subjects did not have surgery. | -1.396 (4.575)
  Lumbar cobb angle change at 1 month: number analyzed (Participants) | 63 | 12 | 36
  Lumbar cobb angle change at 1 month | 0.626 (7.075) | 5.661 (10.117) | 0.839 (5.336)
  Lumbar cobb angle change at 12 months: number analyzed (Participants) | 37 | 6 | 27
  Lumbar cobb angle change at 12 months | 1.232 (7.785) | -1.412 (3.634) | 2.057 (13.535)
  Local cobb angle of T5-L1 at baseline: number analyzed (Participants) | 49 | 9 | 31
  Local cobb angle of T5-L1 at baseline | 22.914 (12.720) | 23.519 (11.363) | 23.847 (15.945)
  Local cobb angle of T5-L1 change at post-op: number analyzed (Participants) | 49 | 23 | 31
  Local cobb angle of T5-L1 change at post-op | -0.506 (4.231) | NA (NA) — Subjects did not have surgery. | -2.080 (5.311)
  Local cobb angle of T5-L1 change at 1 month: number analyzed (Participants) | 45 | 9 | 30
  Local cobb angle of T5-L1 change at 1 month | 1.126 (5.639) | 0.357 (7.731) | -0.746 (5.230)
  Local cobb angle of T5-L1 change at 12 months: number analyzed (Participants) | 29 | 2 | 24
  Local cobb angle of T5-L1 change at 12 months | 1.550 (5.525) | 1.638 (1.998) | -1.333 (4.781)
  Local cobb angle of L2-L4 at baseline: number analyzed (Participants) | 24 | 6 | 16
  Local cobb angle of L2-L4 at baseline | -7.715 (15.470) | -6.581 (9.957) | -6.945 (14.496)
  Local cobb angle of L2-L4 change at post-op: number analyzed (Participants) | 24 | 23 | 16
  Local cobb angle of L2-L4 change at post-op | -1.834 (7.886) | NA (NA) — Subjects did not have surgery. | -0.610 (4.094)
  Local cobb angle of L2-L4 change at 1 month: number analyzed (Participants) | 23 | 6 | 16
  Local cobb angle of L2-L4 change at 1 month | 0.117 (5.694) | -0.105 (5.106) | -0.770 (3.376)
  Local cobb angle of L2-L4 change at 12 months: number analyzed (Participants) | 15 | 3 | 13
  Local cobb angle of L2-L4 change at 12 months | 0.005 (4.925) | -0.346 (3.197) | -1.157 (3.604)

19. Secondary Outcome: Index Spinal Deformity Change Measured by Index Vertebral Body Height Ratio
Description: Index spinal deformity was measured by Kyphotic angle, local Cobb angle, thoracic and lumbar Cobb angle, and anterior, middle and posterior vertebral body heights for each index VCF. Index Vertebral Body Height Ratio (VBHR) was defined as index vertebra height divided by the average of normal superior and inferior adjacent vertebrae.
Time Frame: Baseline and 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
ratio
  Anterior VBHR at baseline: number analyzed (Participants) | 50 | 37
  Anterior VBHR at baseline | 0.744 (0.228) | 0.734 (0.237)
  Anterior VBHR change at 1 month: number analyzed (Participants) | 39 | 33
  Anterior VBHR change at 1 month | 0.016 (0.123) | -0.027 (0.061)
  Medial VBHR at baseline: number analyzed (Participants) | 50 | 37
  Medial VBHR at baseline | 0.782 (0.193) | 0.776 (0.190)
  Medial VBHR change at 1 month: number analyzed (Participants) | 39 | 33
  Medial VBHR change at 1 month | 0.028 (0.103) | -0.017 (0.068)
  Posterior VBHR at baseline: number analyzed (Participants) | 50 | 37
  Posterior VBHR at baseline | 0.928 (0.101) | 0.934 (0.110)
  Posterior change at 1 month: number analyzed (Participants) | 39 | 33
  Posterior change at 1 month | 0.007 (0.081) | -0.012 (0.058)

20. Secondary Outcome: Index Spinal Deformity Change Measured by Index Vertebral Body Height Ratio
Description: as for outcome 19
Time Frame: Baseline, post-operation, 1 month, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
ratio
  Anterior VBHR at baseline: number analyzed (Participants) | 50 | 9 | 27
  Anterior VBHR at baseline | 0.744 (0.228) | 0.767 (0.254) | 0.741 (0.224)
  Anterior VBHR change at post-op: number analyzed (Participants) | 44 | 23 | 25
  Anterior VBHR change at post-op | 0.060 (0.117) | NA (NA) — Subjects did not have surgery. | 0.024 (0.084)
  Anterior VBHR change at 1 month: number analyzed (Participants) | 39 | 9 | 23
  Anterior VBHR change at 1 month | 0.016 (0.123) | -0.036 (0.054) | 0.006 (0.065)
  Anterior VBHR change at 12 months: number analyzed (Participants) | 22 | 4 | 20
  Anterior VBHR change at 12 months | 0.022 (0.129) | -0.022 (0.072) | 0.039 (0.145)
  Medial VBHR at baseline: number analyzed (Participants) | 50 | 9 | 27
  Medial VBHR at baseline | 0.782 (0.193) | 0.741 (0.239) | 0.800 (0.176)
  Medial VBHR change at post-op: number analyzed (Participants) | 44 | 23 | 25
  Medial VBHR change at post-op | 0.044 (0.099) | NA (NA) — Subjects did not have surgery. | 0.019 (0.075)
  Medial VBHR change at 1 month: number analyzed (Participants) | 39 | 9 | 23
  Medial VBHR change at 1 month | 0.028 (0.103) | -0.031 (0.074) | 0.012 (0.071)
  Medial VBHR change at 12 months: number analyzed (Participants) | 22 | 4 | 20
  Medial VBHR change at 12 months | 0.018 (0.110) | 0.021 (0.117) | 0.049 (0.087)
  Posterior VBHR at baseline: number analyzed (Participants) | 50 | 9 | 27
  Posterior VBHR at baseline | 0.928 (0.101) | 0.899 (0.166) | 0.951 (0.110)
  Posterior VBHR change at post-op: number analyzed (Participants) | 44 | 23 | 25
  Posterior VBHR change at post-op | 0.007 (0.064) | NA (NA) — Subjects did not have surgery. | -0.006 (0.059)
  Posterior VBHR change at 1 month: number analyzed (Participants) | 39 | 9 | 23
  Posterior VBHR change at 1 month | 0.007 (0.081) | -0.022 (0.045) | 0.016 (0.069)
  Posterior VBHR change at 12 months: number analyzed (Participants) | 22 | 4 | 20
  Posterior VBHR change at 12 months | -0.001 (0.077) | -0.026 (0.049) | 0.006 (0.053)

21. Secondary Outcome: Back Pain Analgesics Used
Time Frame: Baseline, 7 days, and 1 month
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
percentage of participants
  Back pain analgesic use at baseline: number analyzed (Participants) | 68 | 60
  Back pain analgesic use at baseline | 96 | 84
  Back pain analgesic use at 7 days: number analyzed (Participants) | 63 | 55
  Back pain analgesic use at 7 days | 82 | 80
  Back pain analgesic use at 1 month: number analyzed (Participants) | 64 | 49
  Back pain analgesic use at 1 month | 60 | 72

22. Secondary Outcome: Back Pain Analgesics Used
Time Frame: Baseline, 7 days, 1 month, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
percentage of participants
  Back pain analgesic use at baseline | 96 | 78 | 87
  Back pain analgesic use at 7 days | 82 | 61 | 68
  Back pain analgesic use at 1 month | 60 | 39 | 66
  Back pain analgesic use at 3 months | 43 | 30 | 58
  Back pain analgesic use at 6 months | 40 | 22 | 39
  Back pain analgesic use at 12 months | 19 | 13 | 26

23. Secondary Outcome: Change in Neurology Status From Baseline (Motor Strength)
Description: The neurological examination included motor strength, sensory examination, reflexes below the level of the most cephalad index vertebral body fracture, and the presence of radicular pain. Evaluation criteria of motor strength (scored 0-5) for rectus abdominis, hip extensors and flexors, knee extensors and flexors, and foot plantar and dorsiflexors as following:
  absent voluntary contraction = 0, contractions unable to move joint = 1, movement with gravity eliminated = 2, movement against gravity = 3, movement against resistance = 4, full strength = 5
Time Frame: 1 month
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
percentage of participants
  Improved at 1 month | 8.8 | 3.3
  Unchanged at 1 month | 84 | 74
  Worsened at 1 month | 1.5 | 3.3

24. Secondary Outcome: Change in Neurology Status From Baseline (Motor Strength)-Per Protocol
Description: as for outcome 23
Time Frame: 1 month, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
percentage of participants
  Improved at 1 month | 8.8 | 8.7 | 2.6
  Unchanged at 1 month | 84 | 39 | 92
  Worsened at in month | 1.5 | 4.3 | 2.6
  Improved at 3 months | 7.4 | 4.3 | 7.9
  Unchanged at 3 months | 68 | 35 | 84
  Worsened at 3 months | 2.9 | 4.3 | 2.6
  Improved at 6 months | 5.9 | 4.3 | 11
  Unchanged at 6 months | 62 | 30 | 68
  Worsened at 6 months | 4.4 | 0.0 | 7.9
  Improved at 12 months | 2.9 | 4.3 | 5.3
  Unchanged at 12 months | 53 | 22 | 66
  Worsened at 12 months | 2.9 | 0.0 | 0.0

25. Secondary Outcome: Change in Neurological Status From Baseline (Sensory Examination)
Description: The neurological examination included motor strength, sensory examination, reflexes below the level of the most cephalad index vertebral body fracture, and the presence of radicular pain. For sensory examination, the Investigator assessed sensory status at baseline and a change from baseline beginning with the most cephalad index level treated through L5.
Time Frame: 1 month
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
percentage of participants
  Improved | 2.9 | 1.6
  Unchanged | 91 | 79
  Worsened | 0.0 | 0.0

26. Secondary Outcome: Change in Neurological Status From Baseline (Sensory Examination)
Description: as for outcome 25
Time Frame: 1 months, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
percentage of participants
  Improved at 1 month | 2.9 | 0.0 | 2.6
  Unchanged at 1 month | 91 | 52 | 95
  Worsened at 1 month | 0.0 | 0.0 | 0.0
  Improved at 3 months | 1.5 | 0.0 | 2.6
  Unchanged at 3 months | 78 | 43 | 92
  Worsened at 3 months | 0.0 | 0.0 | 0.0
  Improved at 6 months | 0.0 | 0.0 | 2.6
  Unchanged at 6 months | 71 | 35 | 84
  Worsened at 6 months | 1.5 | 0.0 | 0.0
  Improved at 12 months | 1.5 | 4.3 | 0.0
  Unchanged at 12 months | 57 | 22 | 66
  Worsened at 12 months | 0.0 | 0.0 | 5.3

27. Secondary Outcome: Change in Neurological Status From Baseline (Reflex Strength)
Description: The neurological examination included motor strength, sensory examination, reflexes below the level of the most cephalad index vertebral body fracture, and the presence of radicular pain. Evaluation criteria of reflexes (scored 0-3) for patellar and Achilles reflexes as following:
  absent = 0, hypoactive = 1, normal = 2, brisk or clonus = 3
Time Frame: 1 month
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
percentage of participants
  Improved | 7.4 | 8.2
  Unchanged | 85 | 69
  Worsened | 1.5 | 3.3

28. Secondary Outcome: Change in Neurological Status From Baseline (Reflex Strength)
Description: as for outcome 27
Time Frame: 1 months, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
percentage of participants
  Improved at 1 month | 7.4 | 4.3 | 5.3
  Unchanged at 1 month | 85 | 43 | 82
  Worsened at 1 month | 1.5 | 4.3 | 11.0
  Improved at 3 months | 2.9 | 4.3 | 2.6
  Unchanged at 3 months | 74 | 39 | 82
  Worsened at 3 months | 2.9 | 0.0 | 11.0
  Improved at 6 months | 5.9 | 0.0 | 7.9
  Unchanged at 6 months | 65 | 35 | 71
  Worsened at 6 months | 1.5 | 0.0 | 7.9
  Improved at 12 months | 2.9 | 0.0 | 7.9
  Unchanged at 12 months | 53 | 26 | 63
  Worsened at 12 months | 2.9 | 0.0 | 0.0

29. Secondary Outcome: Change in Neurological Status From Baseline (Limb Strength)
Description: The neurological examination included motor strength, sensory examination, reflexes below the level of the most cephalad index vertebral body fracture, and the presence of radicular pain. Radicular lower limb pain was assessed the presence of paresthesia, weakness, and/or painful straight leg raising (SLR).
Time Frame: 1 month
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 68 | 61
percentage of participants
  Improved | 12 | 4.9
  Unchanged | 81 | 67
  Worsened | 1.5 | 8.2

30. Secondary Outcome: Change in Neurological Status From Baseline (Limb Strength)
Description: as for outcome 29
Time Frame: 1 months, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
percentage of participants
  Improved at 1 month | 12 | 0.0 | 16
  Unchanged at 1 month | 81 | 48 | 82
  Worsened at 1 month | 1.5 | 4.3 | 0.0
  Improved at 3 months | 4.4 | 0.0 | 13
  Unchanged at 3 months | 71 | 39 | 79
  Worsened at 3 months | 4.4 | 4.3 | 2.6
  Improved at 6 months | 7.4 | 0.0 | 13
  Unchanged at 6 months | 63 | 30 | 71
  Worsened at 6 months | 1.5 | 4.3 | 2.6
  Improved at 12 months | 4.4 | 4.3 | 11
  Unchanged at 12 months | 51 | 22 | 58
  Worsened at 12 months | 2.9 | 0.0 | 2.6

31. Secondary Outcome: Rate of Study Treatment-related Adverse Events Within 30 Days of Baseline
Description: The study treatment-related AEs were defined as follows:
  1. Related defined as the AE had a direct relationship to a Sponsor medical device used in the study patient.
  2. Possibly related defined as the AE may have had a relationship to a Sponsor medical device but an alternative cause may be equally or less likely associated.
  3. Unrelated defined as the AE was due to the underlying indication or disease state or to concomitant medication or therapy not related to any Sponsor device.
  4. Unknown defined as the relationship of the AE to a Sponsor device could not be determined.
Time Frame: 1 month
Population: All of the randomized subjects were included in safety population analysis.
Measure: Number; unit: percentage of participants
Groups:
- Balloon Kyphoplasty: The subjects were randomized to the Balloon Kyphoplasty.
- Non Surgical Management: The subjects were randomized to NSM.
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 70 | 64
percentage of participants
  Unrelated | 33 | 30
  Possibly related | 1.4 | 0
  Related | 4.3 | 0
  Unknown | 2.9 | 0

32. Secondary Outcome: Rate of Study Treatment-related Adverse Events Till Study Completion
Description: as for outcome 31
Time Frame: 12 months
Population: All of randomized subjects were included in safety population analysis.
Measure: Number; unit: percentage of participants
Groups:
- Balloon Kyphoplasty: The subjects were randomized to Balloon Kyphoplasty.
- Non Surgical Management: The subjects were randomized to NSM without crossing over.
- Crossover (AEs Collected Before BKP); Crossover-(AEs Collected After BKP): Subjects in this group were randomized to NSM, then, crossed over to Balloon Kyphoplasty after completion of the 1-month evaluation in NSM group.
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover (AEs Collected Before BKP) | Crossover-(AEs Collected After BKP)
Number analyzed (Participants) | 70 | 26 | 38 | 38
percentage of participants
  Unrelated | 77 | 50 | 37 | 79
  Possibly related | 1.4 | 0 | 0 | 2.6
  Related | 4.3 | 0 | 0 | 2.6
  Unknown | 10 | 0 | 0 | 7.9

33. Secondary Outcome: Rate of Subsequent Vertebral Body Fractures
Time Frame: 1 month
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Number analyzed (Participants) | 62 | 47
percentage of participants | 19.6 | 17.0

34. Secondary Outcome: Rate of Subsequent Vertebral Body Fractures
Description: Based on patients with at least 7 analyzable vertebrae.
Time Frame: 1 month and 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Kyphoplasty | Non Surgical Management | Crossover
Number analyzed (Participants) | 68 | 23 | 38
percentage of participants
  1 month: number analyzed (Participants) | 62 | 13 | 34
  1 month | 19.4 | 23.1 | 11.8
  12 months: number analyzed (Participants) | 38 | 6 | 27
  12 months | 13.2 | 0.0 | 7.4

ADVERSE EVENTS:
Time Frame: Adverse Events within 30 Days of treatment
Groups:
- Balloon Kyphoplasty: The subjects assigned to this group will undergo the treatment with Balloon kyphoplasty for their painful VCFs.
Arm/Group | Balloon Kyphoplasty | Non Surgical Management
Serious Adverse Events (participants affected / at risk) | 15/70 | 11/64
Other Adverse Events (participants affected / at risk) | 16/70 | 11/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Kyphoplasty (N=70) | Non Surgical Management (N=64)
Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) — Resulted in death
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — Occurred prior to planned surgery and resulted in death
Gastric hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 1 (1) — Event in kyphoplasty group resulted in death
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Post Procedural Myocardial Infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral Fracture (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (4)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Kyphoplasty (N=70) | Non Surgical Management (N=64)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 0 (0) | 1 (1)
Implant Site Extravasation (General disorders) | 2 (2) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Device Breakage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Event was asymptomatic
Haemoglobin Decreased (Investigations) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less